CLINICAL TRIAL: NCT02470975
Title: How Families Cope With Child Cancer? A Longitudinal Study on the Role of "We-appraisals" on Child's Health-related Quality of Life
Brief Title: How Family Coping With Child Cancer Affects Child's Quality of Life?
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KLS-3325-02-2014
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Children with newly diagnosed cancer and their parents will be contacted and invited to participate. Upon agreement, children will be interviewed, both parents will fill out questionnaires and be additionally interviewed. Using a 3-wave longitudinal design, mainly self-reported parental we-appraisals and we-disease-appraisals, couple dyadic coping (DC) and parent-child DC during a course of 12 months will be examined. Additionally, during brief separate interviews, the parents' speech will be coded for we-appraisals and expressed emotion regarding the other partner and the child. Findings will provide information on how family variables affect child QoL over 12 months.

DETAILED DESCRIPTION:
Background

Researchers and clinicians alike have been calling for family-oriented and longitudinal research on child cancer (CC). The reason for this is threefold. First, parents are the most influential context on child development. Second, CC can be considered a "we-family disease", that is, a stressor that affects the patient, their parents and the interaction within all family members and subsystems, since they are an interdependent unit. Third, the higher survivals rates and increased chronicity of CC demand an ongoing adaptation from the whole family to the illness-related stress. As such, several studies have found associations between family and child variables during and after cancer treatment, and few studies suggest a causal relationship of family functioning on child adjustment and quality of life (QoL). Nevertheless, (1) which family dimensions related with the process of stress, appraisal and coping with CC, (2) how changes and (3) divergences within those dimensions predict child QoL over time, remain answered. Research on stress and coping in couples has identified two crucial dimensions for better relational and health outcomes that have the potential to provide those answers. "We-Appraisals", which is the process how individuals tend to evaluate what happens to them as a couple, i.e., in a more relational-oriented way ("we" problem) or in a more individual way ("I/you" problem); and Dyadic Coping, i.e., the process how couples cope together with stress. Therefore, the aim to expand and understand these dimensions in the context of families coping with CC.

Aims

Using a three-wave longitudinal design, the investigators aim to examine (1) the role that parental we-appraisals and we-disease appraisals, couple and parent-child dyadic coping have for a child's QoL over time, (2) how these variables change over time and how these changes predict changes in a child's QoL, (3) how congruence or discrepancies within we-appraisals and we-disease-appraisals, couple and parent-child dyadic coping predict changes in child's QoL over time, and (4) how observed parental we-appraisals, partner's and parental ex-pressed emotion predict child' QoL.

Hypothesis

The investigators expect that higher scores on parents' variables will predict positive changes on child QoL during the first 12 months after cancer diagnosis (T2 and T3). The investigators expect that changes and discrepancies within parents' variables over time will predict changes in child QoL at T2 and T3.

Methods

One hundred children with newly diagnosed cancer and their mothers and fathers will be recruited from the University Children's Hospitals in Zurich and Berne and assessed three times during 12 months. The children will be interviewed at all time points. The parents will complete several paper-pencil questionnaires assessing the variables of interest and will be interviewed at T2 (6 months) and T3 (1 year). Latent change score models with three factors (i.e. mother, father, child) and multilevel analysis will be used to test our hypothesis.

Relevance

By providing precursor information about the role that key family dimensions play on explaining better child QoL over time, this study will enable health-care professionals to know which family resources and members should be targeted during cancer treatment, improve interventions and, ultimately, to improve child QoL.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 and 17 years old diagnosed with cancer (4-6 weeks) as listed on the Swiss Cancer Registry
* Parents of children recently diagnosed with child cancer
* Caregiver parent living together with another partner in a committed relationship for at least one year.

Exclusion Criteria:

* Ill children with pre-existing severe cognitive and physical disability (physician's rating)
* Ill children with single parents

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with newly diagnosed cancer and their parents
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Child quality of life | Three time points in a 12- months trajectory: 4/6 weeks after cancer diagnosis (T1), 6 months after diagnosis 1 (T2), and 12 months after diagnosis (T3)
  Interview based on the DISABKIDS Chronic Generic Measure long version (DCGM-37) (Ravens-Sieberer et al., 2007)

SECONDARY OUTCOMES:
Child posttraumatic stress disorder | Three time points in a 12- months trajectory: 4/6 weeks after cancer diagnosis (T1), 6 months after diagnosis 1 (T2), and 12 months after diagnosis (T3)
  Interview based on the University of California Los Angeles Child PTSD Reaction Index (Pynoos & Steinberg, 2013, German Version Landolt, 2014)
Parental psychological adjustment | Three time points in a 12- months trajectory: 4/6 weeks after cancer diagnosis (T1), 6 months after diagnosis 1 (T2), and 12 months after diagnosis (T3)
  Measured by the Symptom-Checklist-27 (SCL-27; Hardt, Egle, Kappis, Hessel, & Brähler, 2004)
Parental posttraumatic stress disorder | Three time points in a 12- months trajectory: 4/6 weeks after cancer diagnosis (T1), 6 months after diagnosis 1 (T2), and 12 months after diagnosis (T3)
  Measured by the Posttraumatic Diagnostic Scale (PDS, German version: Elbert et al., 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Landolt, PhD, Principal Investigator — University Children's Hospital of Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Principal Investigator web-site — http://www.psychology.uzh.ch/chairs/gespsy.html